CLINICAL TRIAL: NCT04816942
Title: Clinical Efficacy of Early Administration of Convalescent Plasma Among COVID-19 Cases in Egypt
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ministry of Health and Population, Egypt (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-2020/13
Record Dates: First submitted 2021-02-12; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Convalescent Plasma; Covid19; Immunoglobulins; Plasma; Egypt
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Convalescent Plasma (Experimental): Patients receiving Two units of ABO compatible COVID-19 convalescent plasma will be administered.P
  Interventions: Biological: Convalescent Plasma

INTERVENTIONS:
Biological: Convalescent Plasma — Two units of ABO compatible COVID-19 convalescent plasma will be administered.

SUMMARY:
One investigational treatment being explored for COVID-19 is the use of convalescent plasma collected from individuals who have recovered from COVID-19 (Refs. 1-4). Convalescent plasma that contains antibodies to severe acute respiratory syndrome coronavirus 2 or SARSCoV-2 (the virus that causes COVID-19) is being studied for administration to patients with COVID-19. Use of convalescent plasma has been studied in outbreaks of other respiratory infections, including the 2003 SARS-CoV-1 epidemic, the 2009-2010 H1N1 influenza virus pandemic, and the 2012 MERS-CoV epidemic (Refs. 5-7).

Although promising, convalescent plasma has not yet been shown to be safe and effective as a treatment for COVID-19. Therefore, it is important to study the safety and efficacy of COVID19 convalescent plasma in clinical trials. This guidance provides recommendations to health care providers and investigators on the administration and study of investigational convalescent plasma collected from individuals who have recovered from COVID-19 (COVID-19 convalescent plasma) during the public health emergency. This guidance also provides recommendations to blood establishments on the collection of COVID-19 convalescent plasma..

DETAILED DESCRIPTION:
laboratory-confirmed patients using qRT-PCR will be enrolled in the study. Eligibility criteria for recipients are ; laboratory-confirmed SARS-CoV-2, Severe or immediately life-threatening. Severe disease defined as one or more of the following; shortness of breath( dyspnoea), respiratory frequency≥ 30/min, blood oxygen saturation ≤93%, a partial pressure of arterial oxygen to fraction of inspired oxygen ratio <300, and lung infiltrates >50% within 24-48 hours. While a life-threatening disease is defined as one or more of the following; respiratory failure, need for mechanical ventilation, septic shock and multiple organ dysfunction or failure.

Intervention: All patients included in the study provided will be administered with two plasma units (each unit is 200cc).

Primary measure is the degree of clinical improvement among the COVID-19 patients who receive CPT within seven days as compared with the patients who receive after seven days. Case Fatality will be assessed among the enrolled cases

ELIGIBILITY:
Inclusion Criteria:

Laboratory confirmed COVID-19. Severe or immediately life-threatening COVID-19,

Exclusion Criteria Not fitting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
COVID-19 Cure rate | 30 days
  Primary measure was the degree of clinical improvement among the COVID-19 patients who received CPT within seven days as compared with the patients who received after seven days

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No